CLINICAL TRIAL: NCT02383225
Title: Culturally Grounded Early Substance Use Prevention for American Indian Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 12-1641
Record Dates: First submitted 2014-12-30; First posted 2015-03-09 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Substance Use
Keywords: American Indian; Adolescent; Prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Condition A (Experimental): Substance use resistance skills; no Lakota language enhancement, no FaceBook supplement
  Interventions: Behavioral: Substance Use Resistance Skills
- Condition B (Experimental): FaceBook supplement; no Lakota language enhancement; no Substance Use resistance skills
  Interventions: Behavioral: Facebook Supplement
- Condition C (Experimental): Lakota language enhancement; no FaceBook supplement; no Substance Use resistance skills
  Interventions: Behavioral: Lakota Language enhancement
- Condition D (Experimental): Lakota language enhancement; FaceBook supplement; Substance Use resistance skills
  Interventions: Behavioral: Lakota Language enhancement; Behavioral: Facebook Supplement; Behavioral: Substance Use Resistance Skills

INTERVENTIONS:
Behavioral: Lakota Language enhancement — This intervention component includes more extensive adaptation for Lakota families, focusing on use of Lakota language specifically around relationship/kinship terms. Study arms without this component will include the same adapted intervention but with use of English language rather than Lakota.
  Arms: Condition C; Condition D
Behavioral: Facebook Supplement — This intervention component includes a social media supplement to engage families outside of weekly intervention sessions and will include postings and polls for participating parents/other caregivers to complete between sessions.
  Arms: Condition B; Condition D
Behavioral: Substance Use Resistance Skills — This intervention component consists of the original substance use resistance skills training from the Iowa Strengthening Families Program for Parents and Youth 10-14; arms without this component will include a session on healthy eating and exercise (attention control).
  Arms: Condition A; Condition D

SUMMARY:
This study involves adaptation, implementation, and rigorous evaluation of a family-based program designed to prevent early initiation of substance use on a Northern Plains Indian reservation. The program, Thiwáhe Gluwáš'akapi, is a cultural adaptation of the Iowa Strengthening Families Program for Parents and Youth 10-14. Youth and their parents/caregivers will participate in weekly group sessions for 7 weeks and complete pre- and post-intervention surveys assessing a variety of risk and protective factors and youth outcomes. The evaluation design will allow the assessment of the effectiveness of different components within the program.

DETAILED DESCRIPTION:
Feasibility Pilot

A feasibility pilot for the Thiwáhe Gluwáš'akapi (TG) program will be conducted in the Spring of 2015. In the pilot, the intervention will be delivered to two groups of youth and families and the implementation process will be carefully evaluated to determine what works well and where further adaptation of the intervention or the study procedures may be necessary. Particular attention will be paid to retention of families and, if possible, any who drop out will be interviewed to understand barriers to participation.

As with the intervention evaluation itself (see below) youth aged 10-14 will be recruited to participate, along with their parents and/or other adults (up to 3 adults per child) who are actively involved in raising them (e.g., grandparents, aunts, uncles). Pilot groups will be conducted in each of two different communities on the reservation.

Once the feasibility pilot is complete, the intervention will be finalized for efficacy evaluation. Tasks for this phase will include refining the manual for the intervention and further developing training materials for interventionists.

Implementation/Component Evaluation

The formal evaluation of TG will begin in the fall of 2015 and will utilize the principles of Multiphase Optimization Strategy (MOST; Collins et al., 2009) for intervention development and a fractional factorial design to evaluate the relative effectiveness of different components within the intervention. Three components will be evaluated: (1) A Lakota language enhancement (Lakota), (2) a Facebook social media enhancement (FB), and (3) substance use resistance skill content (SU). A total of 24 intervention groups will be randomly assigned to one of 4 MOST design conditions, with the content of each condition determined using SAS PROC FACTEX, as recommended by Collins, et al, 2009. All 4 conditions will consist of the basic TG program, each supplemented by one or more of 3 components designated above: Condition A will include the substance use resistance content (SU; no Lakota or FB); Condition B will include the FB social media supplement (FB; no Lakota or SU); Condition C will include the Lakota language enhancement (Lakota; no FB or SU); and Condition D will include all three components (Lakota + FB + SU).

A cumulative evidence design will be utilized, with the intervention implemented in 5 cohorts across 3 years. The intervention will be delivered to 4 groups (8 families each) in Cohort 1 in the fall of 2015. Additional cohorts will receive the intervention each fall and spring through 2017 as follows: Cohort 2, Spring 2016, 4 groups; Cohort 3, Fall 2016, 6 groups; Cohort 4, Spring 2017, 6 groups; and Cohort 5, Fall 2017, 4 groups. Thus, by the end of 2017, 24 intervention groups (each 8 families, total of 192 families) will have participated in the TG program. Cohorts will be randomly assigned to the 4 MOST design conditions in order to control for potential order of implementation effects.

Power analysis

Power analyses suggest that this design will result in adequate power (>.80) to detect a small effect (d=.15) with 48 families per condition; for the 4 conditions in the design, this will require a total of 192 families (not including 16 pilot families). TG, following Iowa Strengthening Families Program (ISFP) recommendations, will be delivered in family groups of 8 families each; thus, in order to involve 192 families, we plan a total of 24 intervention groups, with 6 in each the 4 experimental conditions. Each component targeted for evaluation will be implemented in 2 of the 4 conditions (see conditions A-B above), and estimates of each effect will thus be based on marginal Ns of 96 families. As is standard with MOST designs, there will not be a no-intervention control group nor will there be a group that receives every component. While this is a different approach than an randomized controlled trial (RCT) design, it is a rigorous and optimal approach for identifying the most effective components to include in an intervention. The intervention created using this process will be ready for a standard RCT evaluation, and more likely to be proven effective there.

Implementation evaluation

Fidelity across implementations will be ensured by using a detailed manual of procedures, providing extensive training for interventionists, and using fidelity logs to asses delivery of key session components. The intervention director, a clinical psychologist, will observe sessions periodically and verify the extent to which implementation is occurring with fidelity to the TG program manual.

Efficacy evaluation

The primary impetus for the development and implementation of the TG program is the desire to reduce risk for substance abuse problems among American Indian adolescents by preventing early initiation of substance use. Assessment of the success of the TG program components will hinge on observed impacts on substance use initiation and on the putative mediators of parental self-efficacy, strengthened family relationships, and cultural knowledge and values. Given the short timeline of the outcome evaluations (limited to 6 months post-intervention), effects on mediators are anticipated to stronger than distal effects on behavioral outcomes.

Measures

Measures used to assess study outcomes draw heavily from the investigators' previous research with young American Indian adolescents and their parents, and from previous evaluations of the Iowa Strengthening Families Program for Parents and Youth 10-14. Two instruments will be used to assess an array of outcomes expected to be affected by the TG intervention, along with demographic data: a Parent Survey (for parents and other caregivers participating in the TG program with youth), and a Youth Survey. Both the Parent Survey and Youth Survey will be administered electronically, using tablet computers connected to the Internet, with data uploaded directly. In addition, a Social Network Survey will be administered (either on an electronic tablet or on paper) to participating parents/caregivers; this survey is designed to assess the strength of the connections among participants in the program, both before and after participation in the program. A small number of participants (3-4) in each group assigned to the FaceBook condition will be asked to participate in Exit Interviews (by phone) to ascertain their use of and response to the social media messages provided between TG sessions. Data will also be captured from Facebook, including page visits, posts, and responses to online quizzes. Finally, participants will be asked to complete a Program Evaluation Form (Parent or Youth versions, on paper) at their last TG session, to provide feedback on the program and facilitators.

Data Collection Schedule

Time 1 - One week prior to the first TG session: Parent and Youth surveys (all participants).

Time 2 - First TG session: Social Network Surveys (adults).

Time 3 - One week after last TG session: Parent and Youth Surveys (all participants); Social Network Survey (adults)

Time 4 - Within two weeks after final TG session: FaceBook Exit Interviews (3-4 adult participants in each condition including the FaceBook supplement)

Time 5 - Approximately 6 months after the last TG session: Parent and Youth Surveys (all participants in the first two intervention cohorts)

Analyses

The simplest analyses for the evaluation of the TG program, using the MOST design, will involve analysis of variance (ANOVA), using the fractional factorial design described above, comparing post-intervention values (Time 3 and Time 5) on both mediators and outcomes across conditions (assuming that randomization across conditions will result in roughly equivalent pre-intervention values). Repeated measures ANOVA will also be performed, including both pre- and post-intervention measures, looking for interactions between time and condition. Finally, multivariate ANOVAs will be estimated for groups of outcome variables, to examine patterns of effects across outcomes. For all analyses, the focus will be on effect sizes (rather than significance tests and p values) to compare effect sizes across components to guide decisions about what should be retained in the optimized TG intervention. As noted above, standard errors will be adjusted to account for intraclass correlations and clustering of families within intervention groups. Analyses of the Social Network Measure will focus on assessing density and cohesion at the network level, to address two primary questions: First, do network characteristics at the beginning of the program (pre-existing relationships within intervention groups) modify the effect of the TG intervention within those groups and, second, do network characteristics change over the course of the TG intervention as new relationships are formed and existing relationships changed. Analyses will be conducted using UCINET or similar social network analysis software. Analyses of the Facebook data will be primarily descriptive, examining the frequency with which participants engage with the Facebook page for their TG group by posting comments, or responding to polls or quizzes. Exploratory analyses may be used to examine correlations between group rates of Facebook use and group-level outcomes, such as increased cohesion as measured by the Social Network Analysis. Analyses of Facebook Exit Interviews will be primarily notes-based content analysis and will involve three major stages of analysis: open coding, axial coding, and selective coding.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 10-14 years and their families, with connection to the South Dakota Indian Reservation where the study is being conducted. Families may include parents, extended family, guardians, and others living in the household.

Exclusion Criteria:

* Individuals without a child in the family aged 10-14 will not be allowed to participate.
* Youth who are not between 10 and 14 years of age will not be allowed to participate.

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2013-06-15 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Youth lifetime alcohol use | Baseline (1 week before program start)
  Lifetime prevalence of alcohol use
Youth lifetime alcohol use | Post-intervention (1 week after program conclusion)
  Lifetime prevalence of alcohol use
Youth lifetime alcohol use | Follow-up (6 months after program conclusion)
  Lifetime prevalence of alcohol use
Youth past-month alcohol use | Baseline (1 week before program start)
  Mean frequency of past month alcohol use
Youth past-month alcohol use | Post-intervention (1 week after program conclusion)
  Mean frequency of past month alcohol use
Youth past-month alcohol use | Follow-up (6 months after program conclusion)
  Mean frequency of past month alcohol use
Youth maximum alcohol use in past month | Baseline (1 week before program start)
  Mean maximum quantity of past month alcohol consumption
Youth maximum alcohol use in past month | Post-intervention (1 week after program conclusion)
  Mean maximum quantity of past month alcohol consumption
Youth maximum alcohol use in past month | Follow-up (6 months after program conclusion)
  Mean maximum quantity of past month alcohol consumption
Youth age of first alcohol use | Baseline (1 week before program start)
  Mean age of first alcohol use
Youth age of first alcohol use | Post-intervention (1 week after program conclusion)
  Mean age of first alcohol use
Youth age of first alcohol use | Follow-up (6 months after program conclusion)
  Mean age of first alcohol use
Youth lifetime cigarette use | Baseline (1 week before program start)
  Lifetime prevalence of cigarette use
Youth lifetime cigarette use | Post-intervention (1 week after program conclusion)
  Lifetime prevalence of cigarette use
Youth lifetime cigarette use | Follow-up (6 months after program conclusion)
  Lifetime prevalence of cigarette use
Youth past-month cigarette use | Baseline (1 week before program start)
  Mean frequency of past month cigarette use
Youth past-month cigarette use | Post-intervention (1 week after program conclusion)
  Mean frequency of past month cigarette use
Youth past-month cigarette use | Follow-up (6 months after program conclusion)
  Mean frequency of past month cigarette use
Youth age of first cigarette use | Baseline (1 week before program start)
  Mean age of first cigarette use
Youth age of first cigarette use | Post-intervention (1 week after program conclusion)
  Mean age of first cigarette use
Youth age of first cigarette use | Follow-up (6 months after program conclusion)
  Mean frequency of past month cigarette use
Youth prevalence of smokeless tobacco use | Baseline (1 week before program start)
  Lifetime prevalence of smokeless tobacco use
Youth prevalence of smokeless tobacco use | Post-intervention (1 week after program conclusion)
  Lifetime prevalence of smokeless tobacco use
Youth prevalence of smokeless tobacco use | Follow-up (6 months after program conclusion)
  Lifetime prevalence of smokeless tobacco use
Youth frequency of past-month smokeless tobacco use | Baseline (1 week before program start)
  Mean frequency of past month smokeless tobacco use
Youth frequency of past-month smokeless tobacco use | Post-intervention (1 week after program conclusion)
  Mean frequency of past month smokeless tobacco use
Youth frequency of past-month smokeless tobacco use | Follow-up (6 months after program conclusion)
  Mean frequency of past month smokeless tobacco use
Youth age of first smokeless tobacco use | Baseline (1 week before program start)
  Mean age of first smokeless tobacco use
Youth age of first smokeless tobacco use | Post-intervention (1 week after program conclusion)
  Mean age of first smokeless tobacco use
Youth age of first smokeless tobacco use | Follow-up (6 months after program conclusion)
  Mean age of first smokeless tobacco use
Youth lifetime prevalence of e-cigarette use | Baseline (1 week before program start)
  Lifetime prevalence of e-cigarette use
Youth lifetime prevalence of e-cigarette use | Post-intervention (1 week after program conclusion)
  Lifetime prevalence of e-cigarette use
Youth lifetime prevalence of e-cigarette use | Follow-up (6 months after program conclusion)
  Lifetime prevalence of e-cigarette use
Youth past-month e-cigarette use | Baseline (1 week before program start)
  Mean frequency of past month e-cigarette use
Youth past-month e-cigarette use | Post-intervention (1 week after program conclusion)
  Mean frequency of past month e-cigarette use
Youth past-month e-cigarette use | Follow-up (6 months after program conclusion)
  Mean frequency of past month e-cigarette use
Youth lifetime marijuana use | Baseline (1 week before program start)
  Lifetime prevalence of marijuana use
Youth lifetime marijuana use | Post-intervention (1 week after program conclusion)
  Lifetime prevalence of marijuana use
Youth lifetime marijuana use | Follow-up (6 months after program conclusion)
  Lifetime prevalence of marijuana use
Youth past-month marijuana use | Baseline (1 week before program start)
  Mean frequency of past month marijuana use
Youth past-month marijuana use | Post-intervention (1 week after program conclusion)
  Mean frequency of past month marijuana use
Youth past-month marijuana use | Follow-up (6 months after program conclusion)
  Mean frequency of past month marijuana us
Youth age of first marijuana use | Baseline (1 week before program start)
  Mean age of first marijuana use
Youth age of first marijuana use | Post-intervention (1 week after program conclusion)
  Mean age of first marijuana use
Youth age of first marijuana use | Follow-up (6 months after program conclusion)
  Mean age of first marijuana use
Youth lifetime prevalence of huffing glue/gas | Baseline (1 week before program start)
  Lifetime prevalence of huffing
Youth lifetime prevalence of huffing glue/gas | Post-intervention (1 week after program conclusion)
  Lifetime prevalence of huffing
Youth lifetime prevalence of huffing glue/gas | Follow-up (6 months after program conclusion)
  Lifetime prevalence of huffing
Youth past-month huffing | Baseline (1 week before program start)
  Mean frequency of past month huffing
Youth past-month huffing | Post-intervention (1 week after program conclusion)
  Mean frequency of past month huffing
Youth past-month huffing | Follow-up (6 months after program conclusion)
  Mean frequency of past month huffing
Youth age of first huffing | Baseline (1 week before program start)
  Mean age of first huffing
Youth age of first huffing | Post-intervention (1 week after program conclusion)
  Mean age of first huffing
Youth age of first huffing | Follow-up (6 months after program conclusion)
  Mean age of first huffing

SECONDARY OUTCOMES:
Youth perceived consistency of parental discipline practices | baseline (1 week before program start)
  Mean perceived consistency of parental discipline practices score
Youth perceived consistency of parental discipline practices | post-intervention (1 week after program conclusion)
  Mean perceived consistency of parental discipline practices score
Youth perceived consistency of parental discipline practices | follow-up (6 months after program conclusion)
  Mean perceived consistency of parental discipline practices score
Youth perceived parental standard setting | baseline (1 week before program start)
  Mean perceived parental standard setting score
Youth perceived parental standard setting | post-intervention (1 week after program conclusion)
  Mean perceived parental standard setting score
Youth perceived parental standard setting | follow-up (6 months after program conclusion)
  Mean perceived parental standard setting score
Youth perceived parental monitoring | baseline (1 week before program start)
  Mean perceived parental monitoring score
Youth perceived parental monitoring | post-intervention (1 week after program conclusion)
  Mean perceived parental monitoring score
Youth perceived parental monitoring | follow-up (6 months after program conclusion)
  Mean perceived parental monitoring score
Youth perceived parental positive affect | baseline (1 week before program start)
  Mean perceived parental positive affect score
Youth perceived parental positive affect | post-intervention (1 week after program conclusion)
  Mean perceived parental positive affect score
Youth perceived parental positive affect | follow-up (6 months after program conclusion)
  Mean perceived parental positive affect score
Youth perceived parental approval | baseline (1 week before program start)
  Mean perceived parental approval score
Youth perceived parental approval | post-intervention (1 week after program conclusion)
  Mean perceived parental approval score
Youth perceived parental approval | follow-up (6 months after program conclusion)
  Mean perceived parental approval score
Youth perceived parental negative affect | baseline (1 week before program start)
  Mean perceived parental negative affect score
Youth perceived parental negative affect | post-intervention (1 week after program conclusion)
  Mean perceived parental negative affect score
Youth perceived parental negative affect | follow-up (6 months after program conclusion)
  Mean perceived parental negative affect score
Youth perceived parent-child communication | baseline (1 week before program start)
  Mean perceived parent-child communication score
Youth perceived parent-child communication | post-intervention (1 week after program conclusion)
  Mean perceived parent-child communication score
Youth perceived parent-child communication | follow-up (6 months after program conclusion)
  Mean perceived parent-child communication score
Youth perceived parent-child communication about alcohol and drugs | baseline (1 week before program start)
  Mean perceived parent-child communication about alcohol and drugs score
Youth perceived parent-child communication about alcohol and drugs | post-intervention (1 week after program conclusion)
  Mean perceived parent-child communication about alcohol and drugs score
Youth perceived parent-child communication about alcohol and drugs | follow-up (6 months after program conclusion)
  Mean perceived parent-child communication about alcohol and drugs score
Youth perceived enforcement of family rules | baseline (1 week before program start)
  Mean perceived enforcement of family rules score
Youth perceived enforcement of family rules | post-intervention (1 week after program conclusion); follow-up (6 months after program conclusion)
  Mean perceived enforcement of family rules score
Youth perceived enforcement of family rules | follow-up (6 months after program conclusion)
  Mean perceived enforcement of family rules score
Youth perceived parental autonomy support | baseline (1 week before program start)
  Mean perceived parental autonomy support score
Youth perceived parental autonomy support | post-intervention (1 week after program conclusion); follow-up (6 months after program conclusion)
  Mean perceived parental autonomy support score
Youth perceived parental autonomy support | follow-up (6 months after program conclusion)
  Mean perceived parental autonomy support score
Parent-child shared activities - youth report | baseline (1 week before program start)
  Count of parent-child shared activities
Parent-child shared activities - youth report | post-intervention (1 week after program conclusion)
  Count of parent-child shared activities
Parent-child shared activities - youth report | follow-up (6 months after program conclusion)
  Count of parent-child shared activities
Family cohesion - youth report | baseline (1 week before program start)
  Mean family cohesion score
Family cohesion - youth report | post-intervention (1 week after program conclusion)
  Mean family cohesion score
Family cohesion - youth report | follow-up (6 months after program conclusion)
  Mean family cohesion score
Family conflict resolution - youth report | baseline (1 week before program start)
  Mean family conflict resolution score
Family conflict resolution - youth report | post-intervention (1 week after program conclusion)
  Mean family conflict resolution score
Family conflict resolution - youth report | follow-up (6 months after program conclusion)
  Mean family conflict resolution score
Family expressiveness - youth report | baseline (1 week before program start)
  Mean family expressiveness score
Family expressiveness - youth report | post-intervention (1 week after program conclusion)
  Mean family expressiveness score
Family expressiveness - youth report | follow-up (6 months after program conclusion)
  Mean family expressiveness score
Lakota cultural socialization - youth report | baseline (1 week before program start)
  Mean Lakota cultural socialization score
Lakota cultural socialization - youth report | post-intervention (1 week after program conclusion)
  Mean Lakota cultural socialization score
Lakota cultural socialization - youth report | follow-up (6 months after program conclusion)
  Mean Lakota cultural socialization score
Youth perceived parental disapproval of alcohol, tobacco, and marijuana | baseline (1 week before program start)
  Mean disapproval of alcohol, tobacco, and marijuana score
Youth perceived parental disapproval of alcohol, tobacco, and marijuana | post-intervention (1 week after program conclusion)
  Mean disapproval of alcohol, tobacco, and marijuana score
Youth perceived parental disapproval of alcohol, tobacco, and marijuana | follow-up (6 months after program conclusion)
  Mean disapproval of alcohol, tobacco, and marijuana score
Descriptive norms for alcohol, tobacco, and marijuana - youth report | baseline (1 week before program start)
  Mean descriptive norms for alcohol, tobacco, and marijuana score
Descriptive norms for alcohol, tobacco, and marijuana - youth report | post-intervention (1 week after program conclusion)
  Mean descriptive norms for alcohol, tobacco, and marijuana score
Descriptive norms for alcohol, tobacco, and marijuana - youth report | follow-up (6 months after program conclusion)
  Mean descriptive norms for alcohol, tobacco, and marijuana score
Youth antisocial behavior | baseline (1 week before program start)
  Mean antisocial behavior score
Youth antisocial behavior | post-intervention (1 week after program conclusion)
  Mean antisocial behavior score
Youth antisocial behavior | follow-up (6 months after program conclusion)
  Mean antisocial behavior score
Youth prosocial behavior | baseline (1 week before program start)
  Mean prosocial behavior score
Youth prosocial behavior | post-intervention (1 week after program conclusion)
  Mean prosocial behavior score
Youth prosocial behavior | follow-up (6 months after program conclusion)
  Mean prosocial behavior score
Youth deviant peer influences | baseline (1 week before program start)
  Mean deviant peer influences score
Youth deviant peer influences | post-intervention (1 week after program conclusion)
  Mean deviant peer influences score
Youth deviant peer influences | follow-up (6 months after program conclusion)
  Mean deviant peer influences score
Youth prosocial peer influences | baseline (1 week before program start)
  Mean prosocial peer influences score
Youth prosocial peer influences | post-intervention (1 week after program conclusion)
  Mean prosocial peer influences score
Youth prosocial peer influences | follow-up (6 months after program conclusion)
  Mean prosocial peer influences score
Youth peer resistance skills | baseline (1 week before program start)
  Mean peer resistance skills score
Youth peer resistance skills | post-intervention (1 week after program conclusion)
  Mean peer resistance skills score
Youth peer resistance skills | follow-up (6 months after program conclusion)
  Mean peer resistance skills score
Youth lifetime history of stressful life events | baseline (1 week before program start)
  Count of stressful events
Youth lifetime history of stressful life events | post-intervention (1 week after program conclusion)
  Count of stressful events
Youth lifetime history of stressful life events | follow-up (6 months after program conclusion)
  Count of stressful events
Youth stress management skills | baseline (1 week before program start)
  Mean stress management skills score
Youth stress management skills | post-intervention (1 week after program conclusion)
  Mean stress management skills score
Youth stress management skills | follow-up (6 months after program conclusion)
  Mean stress management skills score
Youth psychological well-being | baseline (1 week before program start)
  Mean psychological well-being score
Youth psychological well-being | post-intervention (1 week after program conclusion)
  Mean psychological well-being score
Youth psychological well-being | follow-up (6 months after program conclusion)
  Mean psychological well-being score
Youth knowledge of Lakota kinship terminology | baseline (1 week before program start)
  Count of correct Lakota kinship terms
Youth knowledge of Lakota kinship terminology | post-intervention (1 week after program conclusion)
  Count of correct Lakota kinship terms
Youth knowledge of Lakota kinship terminology | follow-up (6 months after program conclusion)
  Count of correct Lakota kinship terms
Youth self-esteem | baseline (1 week before program start)
  Mean self-esteem score
Youth self-esteem | post-intervention (1 week after program conclusion)
  Mean self-esteem score
Youth self-esteem | follow-up (6 months after program conclusion)
  Mean self-esteem score
General parent-child communication - parent/guardian report | baseline (1 week before program start)
  Mean general parent-child communication score
General parent-child communication - parent/guardian report | post-intervention (1 week after program conclusion)
  Mean general parent-child communication score
General parent-child communication - parent/guardian report | follow-up (6 months after program conclusion)
  Mean general parent-child communication score
Parent-child communication about family issues - parent/guardian report | baseline (1 week before program start)
  Mean general parent-child communication about family issues score
Parent-child communication about family issues - parent/guardian report | post-intervention (1 week after program conclusion)
  Mean general parent-child communication about family issues score
Parent-child communication about family issues - parent/guardian report | follow-up (6 months after program conclusion)
  Mean general parent-child communication about family issues score
Parent-child communication about alcohol and drugs - parent/guardian report | baseline (1 week before program start)
  Mean parent-child communication about alcohol and drugs score
Parent-child communication about alcohol and drugs - parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parent-child communication about alcohol and drugs score
Parent-child communication about alcohol and drugs - parent/guardian report | follow-up (6 months after program conclusion)
  Mean parent-child communication about alcohol and drugs score
Parent/guardian report of youth behavior | baseline (1 week before program start)
  Mean youth behavior score
Parent/guardian report of youth behavior | post-intervention (1 week after program conclusion)
  Mean youth behavior score
Parent/guardian report of youth behavior | follow-up (6 months after program conclusion)
  Mean youth behavior score
Parent/guardian report parent-child shared activities | baseline (1 week before program start)
  Count of shared activities
Parent/guardian report parent-child shared activities | post-intervention (1 week after program conclusion)
  Count of shared activities
Parent/guardian report parent-child shared activities | follow-up (6 months after program conclusion)
  Count of shared activities
Parental monitoring - parent/guardian report | baseline (1 week before program start)
  Mean parental monitoring score
Parental monitoring - parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parental monitoring score
Parental monitoring - parent/guardian report | follow-up (6 months after program conclusion)
  Mean parental monitoring score
General family rules - parent/guardian report | baseline (1 week before program start)
  Mean family rules score
General family rules - parent/guardian report | post-intervention (1 week after program conclusion)
  Mean family rules score
General family rules - parent/guardian report | follow-up (6 months after program conclusion)
  Mean family rules score
Family rules about substance use - parent/guardian report | baseline (1 week before program start)
  Mean substance use rules score
Family rules about substance use - parent/guardian report | post-intervention (1 week after program conclusion)
  Mean substance use rules score
Family rules about substance use - parent/guardian report | follow-up (6 months after program conclusion)
  Mean substance use rules score
Parent discipline practices | baseline (1 week before program start)
  Mean parent discipline practices score
Parent discipline practices | post-intervention (1 week after program conclusion)
  Mean parent discipline practices score
Parent discipline practices | follow-up (6 months after program conclusion)
  Mean parent discipline practices score
Other household member discipline practices | baseline (1 week before program start)
  Mean other household member discipline practices score
Other household member discipline practices | post-intervention (1 week after program conclusion)
  Mean other household member discipline practices score
Other household member discipline practices | follow-up (6 months after program conclusion)
  Mean other household member discipline practices score
Standard setting | baseline (1 week before program start)
  Mean standard setting score
Standard setting | post-intervention (1 week after program conclusion)
  Mean standard setting score
Standard setting | follow-up (6 months after program conclusion)
  Mean standard setting score
Parent-child conflict, parent/guardian report | baseline (1 week before program start)
  Mean parent-child conflict score
Parent-child conflict, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parent-child conflict score
Parent-child conflict, parent/guardian report | follow-up (6 months after program conclusion)
  Mean parent-child conflict score
Parent support, parent/guardian report | baseline (1 week before program start)
  Mean parent support score
Parent support, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parent support score
Parent support, parent/guardian report | follow-up (6 months after program conclusion)
  Mean parent support score
Parental positive affect, parent/guardian report | baseline (1 week before program start)
  Mean parental positive affect score
Parental positive affect, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parental positive affect score
Parental positive affect, parent/guardian report | follow-up (6 months after program conclusion)
  Mean parental positive affect score
Parental negative affect, parent/guardian report | baseline (1 week before program start)
  Mean parental negative affect score
Parental negative affect, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parental negative affect score
Parental negative affect, parent/guardian report | follow-up (6 months after program conclusion)
  Mean parental negative affect score
Parental anger management, parent/guardian report | baseline (1 week before program start)
  Mean parental anger management score
Parental anger management, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean parental anger management score
Parental anger management, parent/guardian report | follow-up (6 months after program conclusion)
  Mean parental anger management score
Parental self-efficacy | baseline (1 week before program start)
  Mean parental self-efficacy
Parental self-efficacy | post-intervention (1 week after program conclusion)
  Mean parental self-efficacy
Parental self-efficacy | follow-up (6 months after program conclusion)
  Mean parental self-efficacy
Family meetings, parent/guardian report | baseline (1 week before program start)
  Mean family meetings score
Family meetings, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean family meetings score
Family meetings, parent/guardian report | follow-up (6 months after program conclusion)
  Mean family meetings score
Family cohesion, parent/guardian report | baseline (1 week before program start)
  Mean family cohesion score
Family cohesion, parent/guardian report | post-intervention (1 week after program conclusion
  Mean family cohesion score
Family cohesion, parent/guardian report | follow-up (6 months after program conclusion)
  Mean family cohesion score
Family conflict resolution, parent/guardian report | baseline (1 week before program start)
  Mean family conflict resolution score
Family conflict resolution, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean family conflict resolution score
Family conflict resolution, parent/guardian report | follow-up (6 months after program conclusion)
  Mean family conflict resolution score
Family expressiveness, parent/guardian report | baseline (1 week before program start)
  Mean family expressiveness score
Family expressiveness, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean family expressiveness score
Family expressiveness, parent/guardian report | follow-up (6 months after program conclusion)
  Mean family expressiveness score
Lakota cultural socialization, parent/guardian report | baseline (1 week before program start)
  Mean Lakota cultural socialization score
Lakota cultural socialization, parent/guardian report | post-intervention (1 week after program conclusion)
  Mean Lakota cultural socialization score
Lakota cultural socialization, parent/guardian report | follow-up (6 months after program conclusion)
  Mean Lakota cultural socialization score
Lakota parenting practices | baseline (1 week before program start)
  Mean Lakota parenting practices score
Lakota parenting practices | post-intervention (1 week after program conclusion)
  Mean Lakota parenting practices score
Lakota parenting practices | follow-up (6 months after program conclusion)
  Mean Lakota parenting practices score
Knowledge of Lakota kinship terminology | baseline (1 week before program start)
  Count of correct Lakota kinship terms
Knowledge of Lakota kinship terminology | post-intervention (1 week after program conclusion)
  Count of correct Lakota kinship terms
Knowledge of Lakota kinship terminology | follow-up (6 months after program conclusion)
  Count of correct Lakota kinship terms
Parent lifetime alcohol use | baseline (1 week before program start)
  Lifetime prevalence of alcohol use
Parent lifetime alcohol use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of alcohol use
Parent lifetime alcohol use | follow-up (6 months after program conclusion)
  Lifetime prevalence of alcohol use
Parent past month alcohol use | baseline (1 week before program start)
  Mean frequency of past month alcohol use
Parent past month alcohol use | post-intervention (1 week after program conclusion)
  Mean frequency of past month alcohol use
Parent past month alcohol use | follow-up (6 months after program conclusion)
  Mean frequency of past month alcohol use
Parent past month alcohol use quantity | baseline (1 week before program start)
  Mean usual quantity of past month alcohol consumption
Parent past month alcohol use quantity | post-intervention (1 week after program conclusion)
  Mean usual quantity of past month alcohol consumption
Parent past month alcohol use quantity | follow-up (6 months after program conclusion)
  Mean usual quantity of past month alcohol consumption
Parent past month alcohol use maximum quantity | baseline (1 week before program start)
  Mean maximum quantity of past month alcohol consumption
Parent past month alcohol use maximum quantity | post-intervention (1 week after program conclusion)
  Mean maximum quantity of past month alcohol consumption
Parent past month alcohol use maximum quantity | follow-up (6 months after program conclusion)
  Mean maximum quantity of past month alcohol consumption
Parent past month alcohol use usual quantity | baseline (1 week before program start)
  Mean usual quantity of past month alcohol consumption
Parent past month alcohol use usual quantity | post-intervention (1 week after program conclusion)
  Mean usual quantity of past month alcohol consumption
Parent past month alcohol use usual quantity | follow-up (6 months after program conclusion)
  Mean usual quantity of past month alcohol consumption
Parent past month alcohol intoxication frequency | baseline (1 week before program start)
  Mean frequency of past month alcohol intoxication
Parent past month alcohol intoxication frequency | post-intervention (1 week after program conclusion)
  Mean frequency of past month alcohol intoxication
Parent past month alcohol intoxication frequency | follow-up (6 months after program conclusion)
  Mean frequency of past month alcohol intoxication
Parent first age of alcohol use | baseline (1 week before program start)
  Mean age of first alcohol use
Parent first age of alcohol use | post-intervention (1 week after program conclusion)
  Mean age of first alcohol use
Parent first age of alcohol use | follow-up (6 months after program conclusion)
  Mean age of first alcohol use
Parent first age of alcohol intoxication | baseline (1 week before program start)
  Mean age of first alcohol intoxication
Parent first age of alcohol intoxication | post-intervention (1 week after program conclusion)
  Mean age of first alcohol intoxication
Parent first age of alcohol intoxication | follow-up (6 months after program conclusion)
  Mean age of first alcohol intoxication
Parent lifetime cigarette use | baseline (1 week before program start)
  Lifetime prevalence of cigarette use
Parent lifetime cigarette use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of cigarette use
Parent lifetime cigarette use | follow-up (6 months after program conclusion)
  Lifetime prevalence of cigarette use
Parent past month cigarette use | baseline (1 week before program start)
  Mean frequency and quantity of past month cigarette use
Parent past month cigarette use | post-intervention (1 week after program conclusion)
  Mean frequency and quantity of past month cigarette use
Parent past month cigarette use | follow-up (6 months after program conclusion)
  Mean frequency and quantity of past month cigarette use
Parent age of first cigarette use | baseline (1 week before program start)
  Mean age of first cigarette use
Parent age of first cigarette use | post-intervention (1 week after program conclusion)
  Mean age of first cigarette use
Parent age of first cigarette use | follow-up (6 months after program conclusion)
  Mean age of first cigarette use
Parent lifetime smokeless tobacco use | baseline (1 week before program start)
  Lifetime prevalence of smokeless tobacco use
Parent lifetime smokeless tobacco use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of smokeless tobacco use
Parent lifetime smokeless tobacco use | follow-up (6 months after program conclusion)
  Lifetime prevalence of smokeless tobacco use
Parent past month smokeless tobacco use | baseline (1 week before program start)
  Mean frequency and quantity of past month smokeless tobacco use
Parent past month smokeless tobacco use | post-intervention (1 week after program conclusion)
  Mean frequency and quantity of past month smokeless tobacco use
Parent past month smokeless tobacco use | follow-up (6 months after program conclusion)
  Mean frequency and quantity of past month smokeless tobacco use
Parent age of first smokeless tobacco use | baseline (1 week before program start)
  Mean age of first smokeless tobacco use
Parent age of first smokeless tobacco use | post-intervention (1 week after program conclusion)
  Mean age of first smokeless tobacco use
Parent age of first smokeless tobacco use | follow-up (6 months after program conclusion)
  Mean age of first smokeless tobacco use
Parent lifetime e-cigarette use | baseline (1 week before program start)
  Lifetime prevalence of e-cigarette use
Parent lifetime e-cigarette use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of e-cigarette use
Parent lifetime e-cigarette use | follow-up (6 months after program conclusion)
  Lifetime prevalence of e-cigarette use
Parent frequency of past-month e-cigarette use | baseline (1 week before program start)
  Mean frequency of past month e-cigarette use
Parent frequency of past-month e-cigarette use | post-intervention (1 week after program conclusion)
  Mean frequency of past month e-cigarette use
Parent frequency of past-month e-cigarette use | follow-up (6 months after program conclusion)
  Mean frequency of past month e-cigarette use
Parent lifetime marijuana use | baseline (1 week before program start)
  Lifetime prevalence of marijuana use
Parent lifetime marijuana use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of marijuana use
Parent lifetime marijuana use | follow-up (6 months after program conclusion)
  Lifetime prevalence of marijuana use
Parent past-month marijuana use | baseline (1 week before program start)
  Mean frequency of past month marijuana use
Parent past-month marijuana use | post-intervention (1 week after program conclusion)
  Mean frequency of past month marijuana use
Parent past-month marijuana use | follow-up (6 months after program conclusion)
  Mean frequency of past month marijuana use
Parent age of first marijuana use | baseline (1 week before program start)
  Mean age of first marijuana use
Parent age of first marijuana use | post-intervention (1 week after program conclusion)
  Mean age of first marijuana use
Parent age of first marijuana use | follow-up (6 months after program conclusion)
  Mean age of first marijuana use
Parent lifetime huffing | baseline (1 week before program start)
  Lifetime prevalence of huffing/inhalant use
Parent lifetime huffing | post-intervention (1 week after program conclusion)
  Lifetime prevalence of huffing/inhalant use
Parent lifetime huffing | follow-up (6 months after program conclusion)
  Lifetime prevalence of huffing/inhalant use
Parent past month huffing | baseline (1 week before program start)
  Mean frequency of past month huffing/inhalant use
Parent past month huffing | post-intervention (1 week after program conclusion)
  Mean frequency of past month huffing/inhalant use
Parent past month huffing | follow-up (6 months after program conclusion)
  Mean frequency of past month huffing/inhalant use
Parent age of first huffing | baseline (1 week before program start)
  Mean age of first huffing/inhalant use
Parent age of first huffing | post-intervention (1 week after program conclusion)
  Mean age of first huffing/inhalant use
Parent age of first huffing | follow-up (6 months after program conclusion)
  Mean age of first huffing/inhalant use
Parent lifetime use of non-prescription painkillers | baseline (1 week before program start)
  Lifetime prevalence of non-prescription painkiller use
Parent lifetime use of non-prescription painkillers | post-intervention (1 week after program conclusion
  Lifetime prevalence of non-prescription painkiller use
Parent lifetime use of non-prescription painkillers | follow-up (6 months after program conclusion)
  Lifetime prevalence of non-prescription painkiller use
Parent past month non-prescription painkiller use | baseline (1 week before program start)
  Mean frequency of past month non-prescription painkiller use
Parent past month non-prescription painkiller use | post-intervention (1 week after program conclusion)
  Mean frequency of past month non-prescription painkiller use
Parent past month non-prescription painkiller use | follow-up (6 months after program conclusion)
  Mean frequency of past month non-prescription painkiller use
Parent lifetime stimulant use | baseline (1 week before program start)
  Lifetime prevalence of stimulant use
Parent lifetime stimulant use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of stimulant use
Parent lifetime stimulant use | follow-up (6 months after program conclusion)
  Lifetime prevalence of stimulant use
Parent past month stimulant use | baseline (1 week before program start)
  Mean frequency of past month huffing/inhalant use
Parent past month stimulant use | post-intervention (1 week after program conclusion)
  Mean frequency of past month huffing/inhalant use
Parent past month stimulant use | follow-up (6 months after program conclusion)
  Mean frequency of past month huffing/inhalant use
Parent lifetime sedative use | baseline (1 week before program start)
  Lifetime prevalence of sedative use
Parent lifetime sedative use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of sedative use
Parent lifetime sedative use | follow-up (6 months after program conclusion)
  Lifetime prevalence of sedative use
Parent past month sedative use | baseline (1 week before program start)
  Mean frequency of past month sedative use
Parent past month sedative use | post-intervention (1 week after program conclusion)
  Mean frequency of past month sedative use
Parent past month sedative use | follow-up (6 months after program conclusion)
  Mean frequency of past month sedative use
Parent lifetime heroin use | baseline (1 week before program start)
  Lifetime prevalence of heroin use
Parent lifetime heroin use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of heroin use
Parent lifetime heroin use | follow-up (6 months after program conclusion)
  Lifetime prevalence of heroin use
Parent past month heroin use | baseline (1 week before program start)
  Mean frequency of past month heroin use
Parent past month heroin use | post-intervention (1 week after program conclusion)
  Mean frequency of past month heroin use
Parent past month heroin use | follow-up (6 months after program conclusion)
  Mean frequency of past month heroin use
Parent lifetime methamphetamine use | baseline (1 week before program start)
  Lifetime prevalence of methamphetamine use
Parent lifetime methamphetamine use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of methamphetamine use
Parent lifetime methamphetamine use | follow-up (6 months after program conclusion)
  Lifetime prevalence of methamphetamine use
Parent past month methamphetamine use | baseline (1 week before program start)
  Mean frequency of past month methamphetamine use
Parent past month methamphetamine use | post-intervention (1 week after program conclusion)
  Mean frequency of past month methamphetamine use
Parent past month methamphetamine use | follow-up (6 months after program conclusion)
  Mean frequency of past month methamphetamine use
Parent lifetime hallucinogen use | baseline (1 week before program start)
  Lifetime prevalence of hallucinogen use
Parent lifetime hallucinogen use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of hallucinogen use
Parent lifetime hallucinogen use | follow-up (6 months after program conclusion)
  Lifetime prevalence of hallucinogen use
Parent past month hallucinogen use | baseline (1 week before program start)
  Mean frequency of past month hallucinogen use
Parent past month hallucinogen use | post-intervention (1 week after program conclusion)
  Mean frequency of past month hallucinogen use
Parent past month hallucinogen use | follow-up (6 months after program conclusion)
  Mean frequency of past month hallucinogen use
Parent lifetime club drug use | baseline (1 week before program start)
  Lifetime prevalence of club drug use
Parent lifetime club drug use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of club drug use
Parent lifetime club drug use | follow-up (6 months after program conclusion)
  Lifetime prevalence of club drug use
Parent past month club drug use | baseline (1 week before program start)
  Mean frequency of past month club drug use
Parent past month club drug use | post-intervention (1 week after program conclusion)
  Mean frequency of past month club drug use
Parent past month club drug use | follow-up (6 months after program conclusion)
  Mean frequency of past month club drug use
Parent lifetime cocaine/crack use | baseline (1 week before program start)
  Lifetime prevalence of cocaine/crack use
Parent lifetime cocaine/crack use | post-intervention (1 week after program conclusion)
  Lifetime prevalence of cocaine/crack use
Parent lifetime cocaine/crack use | follow-up (6 months after program conclusion)
  Lifetime prevalence of cocaine/crack use
Parent past month cocaine/crack use | baseline (1 week before program start)
  Mean frequency of past month cocaine/crack use
Parent past month cocaine/crack use | follow-up (6 months after program conclusion)
  Mean frequency of past month cocaine/crack use
Parent HIV risk behavior | baseline (1 week before program start)
  Lifetime prevalence of HIV risk behavior
Parent HIV risk behavior | post-intervention (1 week after program conclusion)
  Lifetime prevalence of HIV risk behavior
Parent HIV risk behavior | follow-up (6 months after program conclusion)
  Lifetime prevalence of HIV risk behavior
Parent psychological distress | baseline (1 week before program start)
  Mean psychological distress score
Parent psychological distress | post-intervention (1 week after program conclusion)
  Mean psychological distress score
Parent psychological distress | follow-up (6 months after program conclusion)
  Mean psychological distress score
Parent life satisfaction | baseline (1 week before program start)
  Mean life satisfaction score
Parent life satisfaction | post-intervention (1 week after program conclusion)
  Mean life satisfaction score
Parent life satisfaction | follow-up (6 months after program conclusion)
  Mean life satisfaction score

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Whitesell, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States